CLINICAL TRIAL: NCT03969251
Title: Optimizing Treatment for Alcohol Use Disorder (AUD) Using Targeted Transcranial Magnetic Stimulation
Brief Title: Transcranial Magnetic Stimulation (TMS) Treatment for Alcohol Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nassima Ait-Daoud Tiouririne (Other)
Responsible Party: Sponsor-Investigator, Nassima Ait-Daoud Tiouririne, Associate Professor, Director of UVA Center for Leading Edge Addiction Research, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21193
Record Dates: First submitted 2019-03-27; First posted 2019-05-31 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Alcoholism
Keywords: alcohol; alcohol dependence; addiction; alcohol use disorder
MeSH Terms: conditions — Alcoholism; Behavior, Addictive | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Transcranial Magnetic Stimulation (rTMS) (Experimental): repetitive transcranial magnetic stimulation
  Interventions: Device: Transcranial Magnetic Stimulation (rTMS)
- Sham (SS) (Sham Comparator): repetitive sham rTMS
  Interventions: Device: Sham (SS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (rTMS) — active high frequency repetitive TMS of left Dorsolateral Prefrontal Cortex
  Arms: Transcranial Magnetic Stimulation (rTMS)
Device: Sham (SS) — repetitive sham rTMS
  Arms: Sham (SS)

SUMMARY:
This is a pilot study designed to evaluate the efficacy of High Frequency (HF) repetitive transcranial magnetic stimulation (rTMS) of the left dorsolateral prefrontal cortex (L-DLPFC) at improving cognitive flexibility in recently detoxified individuals with alcohol use disorder (AUD) compared to placebo (Sham rTMS). The total number of subjects requested to be randomized is 20. The investigator will need to screen about 40 subjects to have 20 subjects started on rTMS session at a ratio of 2 screens/1 subject randomized.

DETAILED DESCRIPTION:
This is a randomized double- blind, control study.

To test the hypothesis, the investigator propose a 2 phase design:

Phase 1: 6-week trial comparing the efficacy of active high-frequency (HF) rTMS of L-DLPFC versus sham (SS) rTMS to determine if HF rTMS improves cognitive flexibility in recently detoxified alcoholics Phase 2: at the end of TMS phase, all participants will receive cognitive behavioral therapy (CBT) thus permitting participants with AUD to benefit from cognitive restructuring in CBT, and reduce alcohol cravings and drinking outcomes.

This study will recruit 20 individuals with AUD, comprising of both male and female participants, age 22 years and older interested in alcohol drinking abstinence. Participants will be recruited from the inpatient unit upon discharge after receiving a detoxification treatment and therefore will be abstinent at study entry. Prior to treatment onset and weekly throughout the course of treatment, participants will complete cognitive testing/measures, Wisconsin Card Sorting Task (WCST), Dimensional Change Card Sort Task (DCCST), Barratt Impulsiveness Scale (BIS), Flanker Inhibitory Control and Attention Test (FICAT), and List Sorting Working Memory Test (LSWMT) and self-reported craving measures, Alcohol Craving Questionnaire (ACQ-Now), and Obsessive Compulsive Drinking Scale (OCDS). The drinking timeline follow-back, and adverse events will also be assessed weekly for 8 weeks.

Participant will be randomized to either high frequency (HF) or sham repetitive transcranial magnetic stimulation (SS rTMS), which will be done 5 days per week for 6 weeks. At the end of 6 weeks, all participants will receive weekly CBT for a total of 8 weeks. Participants will return at 2 and 4 weeks for follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Right handed males and females who have given written informed consent.
* Age 22 years and above with a history of alcohol use disorder
* Good physical health
* Have a current diagnosis of alcohol use disorder
* Reports at least 4 "heavy drinking days" on average in the past 30 days.
* Have a BAC by breathalyzer equal to 0.000 when the participants signed the informed consent document
* Six months stability on any psychotropic medications
* Not have any unresolved legal problems that could jeopardize continuation or completion of the study.
* Be able to provide written informed consent, able to understand written and oral instructions in English and be able to complete the questionnaires required by the protocol.

Exclusion Criteria:

Please contact site for additional information.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Wisconsin Card Sorting Test (WCST) | Up to 5 months
  This is a neuropsychological task that measures flexibility in thinking, or "set shifting," during changing reinforcement schedules.
Dimensional Change Card Sort Task (DCCST) | Up to 5 months
  This is a neuropsychological task that measures cognitive flexibility and attention.
Flanker Inhibitory Control and Attention Test (FICAT) | Up to 5 months
  This is a neuropsychological task that measures attention and inhibitory control.
List Sorting Working Memory Test (LSWMT) | Up to 5 months
  This is a neuropsychological task that measures working memory.

SECONDARY OUTCOMES:
Drinks Per Drinking Day | Up to 5 months
  The investigator will use timeline follow-back to capture this drinking outcome.
Percentage of Days of Abstinence | Up to 5 months
  The investigator will use timeline follow-back to capture this drinking outcome.
Percentage of Heavy Drinking Days | Up to 5 months
  The investigator will use timeline follow-back to capture this drinking outcome.
Alcohol Craving Questionnaire (ACQ-NOW) | Up to 5 months
  This is a 47-item self-administered, multidimensional state measure of acute alcohol craving adapted from the Cocaine Craving Questionnaire. It measures the subscales of alcohol craving labeled Emotionality, Purposefulness, Compulsivity, and Expectancy.

CONTACTS AND LOCATIONS:
Overall Officials: Nassima Ait-Daoud TIouririne, M.D., Principal Investigator — University of Virginia
Locations (1):
- UVA Center for Leading Edge Addiction Research, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No